CLINICAL TRIAL: NCT00270959
Title: Early Combined Intervention After Traumatic Injury
Brief Title: Patient-Centered Collaborative Care for Preventing Post-Traumatic Stress Disorder After Traumatic Injury
Acronym: TSOS II
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Douglas Zatzick, Professor, University of Washington
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 24069; R01MH073613 (NIH); DSIR 82-SECE
Record Dates: First submitted 2005-12-28; First posted 2005-12-29 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Stepped collaborative care (combination of behavioral therapy and drug therapy)
  Interventions: Behavioral: Cognitive Behavioral Therapy; Behavioral: Motivational Interviewing; Drug: FDA-Approved Anti-Anxiety Medications
- 2 (Active Comparator): Standard care provided to injured trauma survivors
  Interventions: Behavioral: Standard Care Control

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Behavioral therapy includes standard cognitive behavioral therapy, with an emphasis on behavioral activation. Treatment is administered on the basis of the participants' individual needs and may continue for up to 12 months.
  Other Names: CBT
  Arms: 1
Behavioral: Motivational Interviewing — Motivational interviewing is designed to address alcohol and drug use.
  Other Names: MI
  Arms: 1
Drug: FDA-Approved Anti-Anxiety Medications — Participants assigned to receive the combination therapy may receive one or more of the following medications based on their individual needs: fluoxetine, sertraline, paroxetine, buspirone, propranolol, trazodone, and any of the benzodiazepines. Participants may begin receiving medication immediately or anytime within the 12 months post-injury. Form, dosage, frequency, and duration depend on patient need, but all are prescribed in accordance with standards of care.
  Arms: 1
Behavioral: Standard Care Control — Standard care control includes the usual treatment for injured trauma survivors.
  Other Names: BA
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of patient-centered collaborative care that combines behavioral therapy and drug therapy as compared to usual care in reducing symptoms of post-traumatic stress disorder in people who have survived a traumatic injury.

DETAILED DESCRIPTION:
Approximately 2.5 million people in the U.S. are hospitalized each year having sustained injuries during a traumatic event. Injured trauma survivors are at high risk for developing post-traumatic stress disorder (PTSD) and other related conditions. In addition, many of these people experience several physical, financial, social, legal, and medical problems over the course of the year following the trauma. Effective interventions to prevent or remedy these issues have yet to be developed for individuals who undergo inpatient surgery following a traumatic injury and who then continue with outpatient treatment and community rehabilitation. This study will evaluate the effectiveness of patient-centered collaborative care that combines behavioral therapy and drug therapy as compared to usual care in reducing symptoms of PTSD and substance use. The study will also assess the intervention's effectiveness in increasing participants' general functioning and satisfaction with their care post-injury.

Participants in this open label study will be randomly assigned to receive either the standard care provided to injured trauma survivors or a combination of behavioral therapy and drug therapy. Participants assigned to receive the combination therapy may receive one or more of the following medications based on their individual needs: fluoxetine; sertraline; paroxetine; buspirone; propranolol; trazodone; and any of the benzodiazepines. Participants may begin receiving medication immediately or anytime within the 12 months post-injury. Behavioral therapy will also be administered on the basis of the participants' individual needs and may continue for up to 12 months. Participants will also take part in motivational interviews, the first of which will be conducted upon study entry in the hospital ward. Subsequent interviews will be conducted over the phone at Months 1, 3, 6, 9, and 12. Participants will be required to report to the study site only for the initial baseline visit. Outcome measures will include PTSD severity ratings, frequency of substance use, and general functioning reports.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Admitted to Harborview Medical Center with injuries sufficiently severe to require inpatient admission
* Experienced a traumatic injury
* Exhibits symptoms of PTSD while in the hospital ward

Exclusion Criteria:

* History of head, spinal, or other injury that may prevent participation in the ward interview
* Requires immediate intervention due to conditions such as self-inflicted injury, active psychosis, or active mania
* Currently incarcerated
* Likely to face criminal charges
* Lives more than 50-100 miles from Harborview Medical Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2006-06; Primary Completion 2010-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
PTSD ratings | Measured at Year 1
Substance use | Measured at Year 1
General functioning reports | Measured at Year 1

SECONDARY OUTCOMES:
Increased satisfaction with global care | Measured at Year 1
Injury relapse | Measured at Year 5
Work, disability, and legal outcomes | Measured at Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Douglas F. Zatzick, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Zatzick D, Roy-Byrne P, Russo J, Rivara F, Droesch R, Wagner A, Dunn C, Jurkovich G, Uehara E, Katon W. A randomized effectiveness trial of stepped collaborative care for acutely injured trauma survivors. Arch Gen Psychiatry. 2004 May;61(5):498-506. doi: 10.1001/archpsyc.61.5.498. PMID 15123495
- [Background] Zatzick DF, Rivara FP, Nathens AB, Jurkovich GJ, Wang J, Fan MY, Russo J, Salkever DS, Mackenzie EJ. A nationwide US study of post-traumatic stress after hospitalization for physical injury. Psychol Med. 2007 Oct;37(10):1469-80. doi: 10.1017/S0033291707000943. Epub 2007 Jun 11. PMID 17559704
- [Background] Zatzick DF, Russo J, Pitman RK, Rivara F, Jurkovich G, Roy-Byrne P. Reevaluating the association between emergency department heart rate and the development of posttraumatic stress disorder: A public health approach. Biol Psychiatry. 2005 Jan 1;57(1):91-5. doi: 10.1016/j.biopsych.2004.10.005. PMID 15607305
- [Derived] Zatzick D, Jurkovich G, Rivara FP, Russo J, Wagner A, Wang J, Dunn C, Lord SP, Petrie M, O'connor SS, Katon W. A randomized stepped care intervention trial targeting posttraumatic stress disorder for surgically hospitalized injury survivors. Ann Surg. 2013 Mar;257(3):390-9. doi: 10.1097/SLA.0b013e31826bc313. PMID 23222034
- See also: Our study is no longer recruiting, if you are seeking care for PSTD from Harborview Medical Center please follow the link above. — http://depts.washington.edu/hcsats/